CLINICAL TRIAL: NCT00426660
Title: A Multicenter, Open Label, Expanded Access Trial Of Maraviroc
Brief Title: Expanded Access Program for Maraviroc At Multiple Centers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: A4001050; 2006-004306-50 (EudraCT Number); EAP (Other: Alias Study Number); NCT02783001 (obsolete NCT alias)
Record Dates: First submitted 2007-01-22; First posted 2007-01-25 (Estimated); Results first posted 2011-10-17 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-05

CONDITIONS: HIV Infections
Keywords: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: maraviroc

INTERVENTIONS:
Drug: maraviroc — The nominal dose for maraviroc is 300 mg twice a day (BID). However, the dosage of maraviroc should be adjusted based on optimal background therapy (OBT) patient is taking. If OBT includes CYP3A4 inhibitor (with or without inducers) maraviroc dose should be 150 mg BID and if OBT includes CYP3A4 inducer (without inhibitors) maraviroc dose should be 600mg BID. If OBT does not include any CYP3A4 inducers or inhibitors maraviroc dose should be 300 mg BID.

SUMMARY:
To provide access to maraviroc to patients who have limited or no therapeutic treatment options and to collect more safety data in a broader patient population.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be failing to achieve adequate virologic suppression on their current regimen and have HIV-1 RNA greater than or equal to 1000 copies/ml, at screening
* Have only R5 HIV-1 at Screening as verified by the Monogram Biosciences Trofile assay
* Minimum age must be 16 years or minimum adult age as determined by local regulatory authorities or directed by local law.

Exclusion Criteria:

* Failed prior treatment with any CCR5 antagonist, in any ongoing CCR5 trial or having previously prematurely discontinued Maraviroc in trials

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1047 (Actual)
Dates: Start 2007-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (360):
- United States (189):
  - The University of Alabama, Birmingham, Alabama
  - Health Services Center, Hobson City, Alabama
  - El Rio, Special Immunology Associates, Tucson, Arizona
  - Health for Life Clinic PLLC, Little Rock, Arkansas
  - Thomas T Jefferson, MD, Little Rock, Arkansas
  - Vista Medical, Beverly Hills, California
  - AHF Research Center, Beverly Hills, California
  - Orange County Center for Special Immunology, Fountain Valley, California
  - Kaiser Permanente, Hayward, California
  - Living Hope Clinical Trials, Long Beach, California
  - AltaMed Health Services Corporation, Los Angeles, California
  - Kaiser Permanente Medical Center, Los Angeles, California
  - Robert Bolan, MD, Los Angeles, California
  - Maternal-Child and Adolescent Clinic of Infectious Diseases and Virology, Los Angeles, California
  - Peter J. Ruane, M.D. Inc., Los Angeles, California
  - Synergy Hematology-Oncology Associates, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Erlmed Corp ABA Lim-Keith Muiltispecialty Clinic Inc., Los Angeles, California
  - Office of Anthony Mills, MD, Los Angeles, California
  - Office of Dr. Salah Bibi, MD, Modesto, California
  - Bonnie V Bock MD, Newport Beach, California
  - Alta Bates Summit Medical Center, Oakland, California
  - Desert Medical Group, Clinical Research Center, Palm Springs, California
  - Riverside Medical Clinic, Riverside, California
  - Fort Sutter Medical Complex, Sacramento, California
  - Sutter Institute for Medical Research, Sacramento, California
  - Sutter Medical Group, Sacramento, California
  - Quest Clinical Research, San Francisco, California
  - Kaiser Permanente Medical Center, San Francisco, California
  - Kaiser Permanente Santa Clara, Santa Clara, California
  - Shared Medical Research Foundation, Tarzana, California
  - Tarzana Treatment Center, Tarzana, California
  - Bipin Bhagat MD Inc., Victorville, California
  - Kaiser Permanente Colorado, Denver, Colorado
  - Kaiser Permanente of Colorado, Denver, Colorado
  - Denver Infectious Disease Consultants, PLLC, Denver, Colorado
  - Kaiser Permanente of Colorado, Lafayette, Colorado
  - Connecticut Health Care Group, Glastonbury, Connecticut
  - Infectious Disease Clinic, Norwich, Connecticut
  - Dupont Circle Physicians Group, Washington D.C., District of Columbia
  - Internal Medicine Associates of Lee County, Bonita Springs, Florida
  - Infectious Disease Research Corp, Boynton Beach, Florida
  - Internal Medicine Associates of Lee County, Cape Coral, Florida
  - Daniel Warner M.D., P.A. Consultive Medicine, Daytona Beach, Florida
  - Northpoint Medical, PA, Fort Lauderdale, Florida
  - Therafirst Medical Centers, Fort Lauderdale, Florida
  - Comprehensive Care Center, Fort Lauderdale, Florida
  - Office of Gary J. Richmond, MD, Fort Lauderdale, Florida
  - Internal Medicine Associates of Lee County, Fort Myers, Florida
  - Sunshine Medical Institute, Hollywood, Florida
  - Osler Medical Inc., Melbourne, Florida
  - Steinhart Medical Associates, Miami, Florida
  - Care Resource, Miami, Florida
  - Office of Albert Canas, MD, Miami Beach, Florida
  - Donald Johnson, MD, North Miami Beach, Florida
  - Wohlfeiler, Piperato & Associates, LLC, North Miami Beach, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Infectious Diseases of Central Florida, Orlando, Florida
  - Associates in Infectious Diseases, Port Saint Lucie, Florida
  - Barry Rodwick, MD, Safety Harbor, Florida
  - Infectious Diseases Associates, Sarasota, Florida
  - University Hepatitis Center at Bach & Godofsky, MD,PA, Sarasota, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Eric Nicholson, M.D., P.A., Tallahassee, Florida
  - University of South Florida, Tampa, Florida
  - University of Sout Florida, Tampa, Florida
  - Midtown Medical Center, Tampa, Florida
  - Donald Watren MD, West Palm Beach, Florida
  - Philip Brachman MD, Atlanta, Georgia
  - Family Health Care of Atlanta, Atlanta, Georgia
  - Midtown West Medical, Atlanta, Georgia
  - Absolute CARE, Atlanta, Georgia
  - Kaiser Permanente, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Infectious Disease Specialists of Atlanta, Decatur, Georgia
  - Kaiser Permanente, Jonesboro, Georgia
  - Infectious Diseases Associates, PC, Riverdale, Georgia
  - Chatham County Health Department, Savannah, Georgia
  - Infectious Disease Consultants, Tucker, Georgia
  - Ruth M. Rothstein CORE Center, Chicago, Illinois
  - Roger Trinh, Chicago, Illinois
  - Northstar Medical Center, Chicago, Illinois
  - Cotton-O'Neil Clinic, Topeka, Kansas
  - Kansas University Internal Medicine Midtown Clinic, Wichita, Kansas
  - Via Christi Research, Inc., Wichita, Kansas
  - Chase Brexton Health Services Inc, Baltimore, Maryland
  - Metro Health Care, Greenbelt, Maryland
  - Dr.'s Alpert, Trinh, and Posorske, Silver Spring, Maryland
  - Tufts - New England Medical Center, Boston, Massachusetts
  - Fenway Community Health, Boston, Massachusetts
  - Community Research Initiative of New England, Boston, Massachusetts
  - Community Research Initiative of New England, Springfield, Massachusetts
  - The Office of Dr. Paul A. Benson, DO, Berkley, Michigan
  - Private Practice (Dr. Gregory Kuldanek), Grand Rapids, Michigan
  - St. John hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Private Practice, Keego Harbor, Michigan
  - MSU Adult Medicine, 10, Lansing, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Nemechek Health Renewal, Kansas City, Missouri
  - Private Practice (Dr. Mark Scheperle), St Louis, Missouri
  - Partnership Health Center, Missoula, Montana
  - CPMC Research Pharmacy, Englewood, New Jersey
  - Leonia Medical Associates, Englewood, New Jersey
  - Center for Infectious Diseaes, Hackensack, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - UMDNJ, Newark, New Jersey
  - University Hospital, Newark, New Jersey
  - Newark Community Health Center, Newark, New Jersey
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - Premier Medical Research Group, Toms River, New Jersey
  - Garden State Infectious Disease Associates, PA, Voorhees Township, New Jersey
  - Upstate Infectious Disease Associates, Albany, New York
  - Woodhull Medical Center, Brooklyn, New York
  - New York Methodist Hospital, Brooklyn, New York
  - NYM Medical Pavilion, Brooklyn, New York
  - Chiu-Bin Hsiao, MD, Buffalo, New York
  - The Office of Dr. Zale P. Bernstein, MD., Buffalo, New York
  - NYHQ, Flushing, New York
  - Schneider Children's Hospital, Great Neck, New York
  - North Shore University Hospital, Department of Infectious Disease, Manhasset, New York
  - Astor Medical Group, LLP, New York, New York
  - Beth Israel Medical Center, New York, New York
  - Paul Bellman, MD, New York, New York
  - Sidney Hillman Family Health Center, New York, New York
  - Ricky Hsu, New York, New York
  - Bellevue Hospital, New York, New York
  - NYU School of Medicine, New York, New York
  - Perion Smith, New York, New York
  - James I Jones Jr, MD, New York, New York
  - Sharon Lewin MD and Michael Rendel MD, New York, New York
  - Lenox Ave Clinic, New York, New York
  - Harlem Medical Associates, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - New York-Presbyterian Hospital, New York, New York
  - Dr. Steven Fine, Rochester, New York
  - Jordon Glaser, MD, Stanton Island, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Allmed Medical and Rehabilitaion of NY, The Bronx, New York
  - Bronx Lebanon Hospital Center, The Bronx, New York
  - ID Associates, Gastonia, North Carolina
  - Rosedale Infectious Diseases, Huntersville, North Carolina
  - Metro Health Systems, Cleveland, Ohio
  - South Dayton Acute Care Consultants Inc., Dayton, Ohio
  - University of Toledo - Health Science Campus, Toledo, Ohio
  - University of Oklahoma - Schusterman Clinic, Tulsa, Oklahoma
  - The Research & Education Group, Portland, Oregon
  - Kaiser Permanente-Northwest Region, Immune Deficiency Clinic, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - RPS Infectious Diseases, West Reading, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - Investigational Drug Services, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Infectious Disease Associates of Memphis, Memphis, Tennessee
  - The Office of Dr. Nicholaos C. Bellos, MD, Dallas, Texas
  - The Office of Dr. Patrick W. Daly, MD., Dallas, Texas
  - The Office of Dr. Susan M. Diamond, MD., Dallas, Texas
  - La Fe CARE Center Clinic, El Paso, Texas
  - Kelly, Allan Rowman MD, Fort Worth, Texas
  - Tarrant County Infectious Disease Associates, Fort Worth, Texas
  - Fernando Garcia, MD, Harlingen, Texas
  - Harris County Hospital District, Houston, Texas
  - Thomas Street Clinic, Houston, Texas
  - Diversified Medical Practices, PA, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - The University of Texas Health Sciences Center at Houston, Houston, Texas
  - Brewton, Gary W MD, Houston, Texas
  - Research Access Network, Houston, Texas
  - The Office of Dr. Gordon E. Crofoot, MD., Houston, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Diagnostic Clinic of Longview, PA, Longview, Texas
  - Dr. James Bromley, San Antonio, Texas
  - Responsive ID Solutions, San Antonio, Texas
  - Clinical Alliance for Research & Education - Infectious Diseases, Annandale, Virginia
  - Infectious Diseases, Arlington, Virginia
  - Infectious Diseases Associates of Central Virginia, Danville, Virginia
  - Infectious Disease Consultants, Fairfax, Virginia
  - Hampton Roads Medical Specialists, Hampton, Virginia
  - Barbara Cassie, Lynchburg, Virginia
  - Crossover Ministry, Richmond, Virginia
  - William F. Ehni, MD, Edmonds, Washington
  - Emerald City Medical Arts, Seattle, Washington
  - Group Health Cooperative, Seattle, Washington
  - The Office of Dr. Daniel R. Coulston, MD, Spokane, Washington
  - The Vancouver Clinic, Inc., P.S., Vancouver, Washington
  - CAMC Memorial Hospital, Charleston, West Virginia
  - Clinical Trials Center, Charleston, West Virginia
  - University Physicians Internal Medicine, Huntington, West Virginia
- Argentina (2):
  - Fundacion Huesped, Departamento de Investigacion Clinica, Buenos Aires
  - FUNCEI, Buenos Aires
- Australia (11):
  - Holdsworth House Medical Practice, Darlinghurst, New South Wales
  - St. Vincent's Hospital, Darlinghurst, New South Wales
  - Albion Street Centre, Surry Hills, New South Wales
  - Westmead Hospital, Wentworthville, New South Wales
  - AIDS Medical Centre, Brisbane, Queensland
  - Infectious Diseases Unit, Herston, Queensland
  - Infectious Diseases Unit, Adelaide, South Australia
  - Melbourne Sexual Health Centre, Carlton, Victoria
  - Northside Clinic, Fitzroy North, Victoria
  - Clinical Research Unit, Infectious Diseases, Melbourne, Victoria
  - Prahran Market Clinic, South Yarra, Victoria
- Austria (3):
  - Allgemeines Krankenhaus Wien, A-1090
  - Landeskrankenhaus Graz West / Abteilung fuer Innere Medizin 1, Graz
  - Sozialmedizinisches Zentrum Baumgartner Hoehe / 2. Interne Lungenabteilung, Vienna
- Belgium (9):
  - Instituut voor Tropische Geneeskunde, Inwendige Geneeskunde, Antwerp
  - Centre Hospitalier Universitaire Saint-Pierre, Maladies Infectieuses, Brussels
  - Hôpital Erasme, Médecine Interne, Brussels
  - Cliniques Universitaires Saint-Luc, Maladies Infectieuses, Brussels
  - Centre Hospitalier Universitaire de Charleroi, Médecine Interne, Charleroi
  - Universitair Ziekenhuis Gent, Inwendige Geneeskunde, Ghent
  - Academisch Ziekenhuis VUB, Jette
  - Universitair Ziekenhuis Gasthuisberg, Inwendige Geneeskunde, Leuven
  - CHU Sart-Tilman, Medecine Interne, Liège
- Canada (8):
  - Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia
  - Hamilton Health Sciences - McMaster University Medical Centre, Hamilton, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Canadian Immunodeficiency Research Collaborative, Toronto, Ontario
  - Clinique médicale l'Actuel, Montreal, Quebec
  - Clinique Medicale du Quartier Latin, Montreal, Quebec
  - CHUM Hôtel-Dieu, Montreal, Quebec
  - Projet L.O.R.I., Montreal, Quebec
- Chile (2):
  - Hospital Clínica Universidad Católica, Santiago, RM
  - Hospital Clínico San Borja Arriarán, Santiago, RM
- Fundación para el Desarrollo de la Lucha contra el SIDA, Barrio Aranjuez, Provincia de San José, Costa Rica
- Instituto Dominicano de Estudios Virologicos, Santo Domingo, Dominican Republic
- France (27):
  - Hopital Sainte Marguerite, Marseille, Cedex 09
  - Hopital Saint Antoine, Paris, Cedex 12
  - Centre Hospitalier Universitaire de Caen, Caen, Cedex
  - Hôpital Saint Jacques, Besançon, France
  - Hopital Gabriel Montpied, Clermont-Ferrand, France
  - CHU Michallon, Grenoble, France
  - Centre Hospitalier Cochin Saint Vincent de Paul, Paris, France
  - Chu Pontchaillou, Service des maladies infectieuses, Rennes, France
  - Hôpital de Purpan, Toulouse, France
  - Hopital Avicenne, Bobigny
  - Hôpital Saint-andré, Bordeaux
  - Hopital Pellegrin - Service des Maladies Infectieuses et Medecine Interne, Bordeaux
  - Hopital La Source, La Source
  - Hopital de Bicêtre, Le Kremlin-Bicêtre
  - Hôpital de la Croix Rousse, Lyon
  - Hopital de l'Hotel-Dieu, Service d'Hepato-Gastroenterologie, Lyon
  - Hopital Gui de Chauliac, Montpellier
  - CHU de Nantes - Hopital Hotel Dieu, Nantes
  - Hopital de l Archet 1, Nice Cedex 3, 06
  - Hôpital de la Pitié Salpétrière, Paris
  - Hopital Europeen George Pompidou, Paris
  - Hopital Bichat-Claude Bernard, Service des Maladies Infectieuses, Paris
  - Hopital Tenon, Service des Maladies Infectieuses, Paris
  - Hopital Saint-Louis, Paris
  - Hôpital Necker-Service des Maladies Infectieuses et Tropicales, Paris
  - CHU de Tourcoing, Tourcoing
  - Hopital Paul Brousse, Villejuif
- Germany (6):
  - Praxisgemeinschaft Bieniek & Cordes, Berlin
  - Universitaetsklinikum Koeln, Klinik I fuer Innere Medizin,, Cologne
  - Universitaetsklinikum Carl Gustav Carus, Klinik und Poliklinik fuer Dermatologie, Dresden
  - Universitaetsklinikum Essen, HIV-Ambulanz, Hautklinik, Essen
  - Gemeinschaftspraxis Dres. Rump und Usadel, Freiburg im Breisgau
  - Medizinische Hochschule Hannover, Klinische Immunologie, Zentrum Innere Medizin, Hanover
- Greece (7):
  - Evagelismos Hospital, Athens, Attica
  - Greek Red Cross Hospital, Athens, Attica
  - General Hospital of Athens G. Gennimatas, Athens
  - Andreas Sygros Hospital, Athens
  - University Hospital of Patras, Pátrai
  - Regional General Hospital Tzaneio, Piraeus
  - AHEPA Hospital, Thessaloniki
- Department of Medicine Queen Elizabeth Hospital, Kowloon, Hong Kong
- India (3):
  - Department of Medicine, St. John's Medical College Hospital, Bangalore, Karnataka
  - Department of HIV Medicine (I D Clinic), Jaslok Hospital & Research Centre, Mumbai, Maharashtra
  - YR Gaitonde Centre for AIDS Research and Education (YRG CARE), Chennai, Tamil Nadu
- Ireland (2):
  - Catherine McAuley Centre, Dublin
  - St. James's Hospital, Dublin
- Italy (24):
  - Universita' degli Studi di Bari, Clinica Malattie Infettive, Policlinico, Bari
  - Unita' Operativa Malattie Infettive, Bologna
  - Istituto di Malattie Infettive e Tropicali, Brescia
  - Unita' Operativa di Malattie Infettive, Catania
  - Presidio Ospedaliero SS Annunziata, Chieti Scalo
  - Arcispedale S. Anna Azienda Ospedaliera Universitaria di Ferrara, Ferrara
  - SOD Malattie Infettive, La Piastra dei Servizi, Florence
  - Unita' Operativa Clinica Malattie Infettive, Dipartimento di Medicina Interna e Malattie Infettive, Genova
  - Fondazione Centro San Raffaele del Monte Tabor, Milan
  - Dipartimento di Scienze Cliniche, Divisione Clinicizzata Malattie Infettive, Milan
  - Clinica Malattie Infettive e Tropicali, Universita' degli Studi di Modena Reggio Emilia, Modena
  - Unita Operativa di Malattie Infettive e Tropicali, Padua
  - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - Reparto di Malattie Infettive, Azienda Sanitaria Locale, Pescara
  - Policlinico Tor Vergata, Divisione Malattie Infettive, Roma
  - IRCCS Lazzaro Spallanzani Istituto Nazionale per la Malattie Infettive, Roma
  - IRCCS Lazzaro Spallanzani Istituto Nazionale per le Malattie Infettive, Roma
  - IRCCS Lazzaro Spallanzani, Istituto Nazionale per le Malattie Infettive, Roma
  - Dipartimento di Malattie Infettive e Tropicali, Universita' di Roma La Sapienza, Roma
  - Universita'Cattolica del Sacro Cuore Policlinico Gemelli, Roma
  - Azienda Ospedaliera San Giovanni Addolorata, Roma
  - Clinica Universitaria di Malattie Infettive, Ospedale Amedeo di Savoia, Torino
  - Uni. Politecnica delle Marche, Ist. Malattie Infettive e Medicina P., Torrette Di Ancona
  - Unita' Operativa di Malattie Infettive, Venezia
- Malaysia (2):
  - Physician Clinic, Kota Bharu, Kelantan
  - Hospital Sungai Buloh, Sungai Buloh, Selangor
- Mexico (3):
  - Antiguo Hospital Civil de Guadalajara "Fray Antonio Alcalde", Guadalajara, Jalisco
  - Hospital Regional Lic. Adolfo Lopez Mateos, Mexico City, Mexico City
  - Instituto Nacional de Ciencias Medicas Y Nutricion Dr Salvador Zubiran, Tlalpan, Mexico Df
- Academisch Ziekenhuis Utrecht, Utrecht, Netherlands
- Portugal (4):
  - Centro Hospitalar de Cascais, Cascais
  - Centro Hospitalar de Lisboa - Zona Central - Hospital Santo António Capuchos, Lisbon
  - Hospital Sta. Maria, Lisbon
  - Hospital São João, Porto
- Puerto Rico (2):
  - Centro Ararat Inc, Ponce, PR
  - HOPE Clinical Research, San Juan
- Romania (4):
  - Spitalul Clinic de Boli Infectioase Constanta, Constanța, Constanța County
  - Spitalul Clinic de Boli Infectioase Sf. Parascheva, Iași, Iaşi
  - Institutul de Boli Infectioase "Prof. Matei Bals", Bucharest, Sector 2
  - Spitalul de Boli Infectioase si Tropicale Victor Babes, Bucharest
- Spain (39):
  - Hospital General Universitario de Alicante, Alicante, Alicante
  - Hospital General Universitario de Elche, Elche, Alicante
  - H. Universitari Germans Trias I Pujol, Badalona, Barcelona
  - Hospital Del Mar, Barcelona, Barcelona
  - Fund. de Gest. Sanitaria de L' Hospital de La Sta. Creu I Sant Pau, Barcelona, Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona, Barcelona
  - Hospital Clinic I Provincial de Barcelona, Barcelona, Barcelona
  - Hospital General de Granollers, Granollers, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital de Basurto, Basurto, Bilbao
  - Hospital Puerta Del Mar, Cadiz, Cadiz
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario Reina Sofia, Córdoba, Cordoba
  - Hospital de Cabueñes, Cabueñes, Gijon
  - Hospital Universitario San Cecilio, Granada, Granada
  - Hospital Universitario Virgen de Las Nieves, Granada, Granada
  - Hospital Clinico Universitario de Santiago de Compostela, Santiago de Compostela, La Coruña
  - Hospital Universitario de La Princesa, Madrid, Madrid
  - Hospital General Gregorio Marañon, Madrid, Madrid
  - Hospital Carlos Iii, Madrid, Madrid
  - Hospital Ramon Y Cajal, Madrid, Madrid
  - Fundacion Jimenez Diaz, Madrid, Madrid
  - Hospital 12 de Octubre, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Complejo Hospitalario Carlos Haya, Málaga, Malaga
  - Hospital Virgen de La Victoria, Málaga, Malaga
  - Hospital Costa Del Sol, Málaga, Malaga
  - Complejo Hospitalario Xeral-Cies, Vigo, Pontevedra
  - Hospital Donostia-Donostia Ospitalea, Donostia / San Sebastian, San Sebastian
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz de Tenerife
  - Hospital Virgen Del Rocio, Seville, Sevilla
  - Complejo Hospitalario Nuestra Señora de Valme, Seville, Sevilla
  - Hospital Universitario Virgen de La Macarena, Seville, Sevilla
  - Hospital de Tortosa Verge de La Cinta, Tortosa, Tarragona
  - Hospital Universitario La Fe, Valencia, Valencia
  - Hospital Clinico Universitario, Valencia, Valencia
  - Consorcio Hospital General Universitario de Valencia, Valencia, Valencia
  - Hospital Arnau de Vilanova, Valencia, Valencia
  - Hospital de Cruces, Barakaldo, Vizcaya
- Universitätsspital Zürich, Zurich, Switzerland
- Department of Infectious Disease, E-Da Hospital, Kaohsiung County, Taiwan
- United Kingdom (7):
  - Brighton and Sussex University Hospitals NHS Trust, The Elton John Centre, Brighton, Sussex
  - North Manchester General Hospital, Crumpsall, Manchester
  - Regional Infectious Diseases Unit, Edinburgh
  - Ian Charleson Centre, London
  - Department of Sexual Health, London
  - St Stephens Research Ltd, London
  - Imperial College, London

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4001050&StudyName=Expanded%20Access%20Program%20for%20Maraviroc%20At%20Multiple%20Centers

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 2584 participants screened, 1047 participants were enrolled in the study.
Groups:
- Maraviroc: Maraviroc 150 milligrams (mg) twice daily (BID), 600 mg BID, or 300 mg BID; dose administered depending on concomitant medications in combination with optimized background therapy (OBT) according to local standard of care.
Period: Overall Study
Arm/Group | Maraviroc
Started | 1047
Treated | 1032
Safety Analysis Set | 1032
Completed | 916
Not Completed | 131
Not completed — Death | 14
Not completed — Adverse Event | 23
Not completed — Insufficient Clinical Response | 22
Not completed — Lost to Follow-up | 15
Not completed — Other | 23
Not completed — Withdrawal by Subject | 18
Not completed — Protocol Violation | 1
Not completed — Enrolled Not Treated | 15

BASELINE CHARACTERISTICS:
Arm/Group | Maraviroc
Number analyzed (Participants) | 1032
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 205
  Male | 827
Baseline Viral Load: Absolute Value [Mean (Standard Deviation); unit: copies/mL] — Human Immunodeficiency Virus (HIV-1) Ribonucleic Acid (RNA) at baseline (BL) (original scale). BL value calculated as average of screening and BL values if both values were within 1 log10 difference. N = number of participants contributing to summary statistic at BL. Viral loads were not available uniformly for all participants enrolled in study.
  copies/mL
    Overall: Absolute (N=979) | 117846.1 (321426.5)
    < 100,000: Absolute (N=729) | 22395.9 (25974.4)
    >= 100,000: Absolute (N=250) | 396179.0 (547142.6)
Baseline Viral Load: Absolute Value [Median (Full Range); unit: copies/mL] — HIV-1 RNA at baseline (BL)(original scale). BL value calculated as average of screening and BL values if both values were within 1 log10 difference. N = number of participants contributing to summary statistic at BL. Viral loads were not available uniformly for all participants enrolled in study.
  copies/mL
    Overall: Absolute (N=979) | 25109.5 [39.0 to 5728492.0]
    < 100,000: Absolute (N=729) | 11028.5 [39.0 to 99643.0]
    >= 100,000: Absolute (N=250) | 234750.0 [100000.0 to 5728492.0]
Baseline Viral Load: Log Scale [Mean (Standard Deviation); unit: log10 copies/mL] — HIV-1 RNA at baseline (BL)(log10 copies/mL). BL value calculated as average of screening and BL values if both values were within 1 log10 difference. N = number of participants contributing to summary statistic at BL. Viral loads were not available uniformly for all participants enrolled in study.
  log10 copies/mL
    Overall: Log Scale (N=979) | 4.259 (1.0182)
    < 100,000: Log Scale (N=729) | 3.859 (0.8517)
    >= 100,000: Log Scale (N=250) | 5.423 (0.3496)
Baseline Viral Load: : Log Scale [Median (Full Range); unit: log10 copies/mL] — HIV-1 RNA at baseline (BL)(log10 copies/mL). BL value calculated as average of screening and BL values if both values were within 1 log10 difference. N = number of participants contributing to summary statistic at BL. Viral loads were not available uniformly for all participants enrolled in study.
  log10 copies/mL
    Overall: Log Scale (N=979) | 4.400 [1.591 to 6.758]
    < 100,000: Log Scale (N=729) | 4.043 [1.591 to 4.998]
    >= 100,000: Log Scale (N=250) | 5.371 [5.000 to 6.758]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Grade 3 and Grade 4 Adverse Events (AE)
Description: AEs as defined by the Division of AIDS (DAIDS) toxicity grading scale: Grade 3 = severe: interrupted usual daily activity and traditionally required systemic drug therapy or other treatment. Grade 4 = very severe: events that were unacceptable and intolerable or were irreversable or caused imminent danger of death. If same participant had more than 1 occurrence in the same preferred term event category, only the most severe (grade 4) occurrence was taken. Treatment-related = investigator assessment of a reasonable possibility that the investigational product caused or contributed to the AE.
Time Frame: Baseline up to Week 144
Population: Safety analysis set: all participants who were randomized and received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 1032
percentage of participants
  Grade 3 AE: all causality | 13.2
  Grade 3 AE: treatment related | 2.4
  Grade 4 AE: all causality | 6.3
  Grade 4 AE: treatment related | 1.6

2. Primary Outcome: Percentage of Participants With Grade 3 Laboratory Abnormalities Without Regards to Baseline Abnormalities
Description: Laboratory abnormalities as defined by the Division of AIDS (DAIDS) toxicity grading scale: Grade 3, Severe =events that interrupted participants usual daily activity and traditionally required systemic drug therapy or other treatment.
Time Frame: Baseline up to Week 144
Population: Safety analysis set. N = number of participants evaluable for laboratory abnormalities (with at least one observation of a laboratory test while on study treatment or during lag time); n = number of participants with at least one observation of given laboratory test while on study treatment or during lag time.
Measure: Number; unit: percentage of participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 1014
percentage of participants
  Alanine aminotransferase (ALT) (n=1013) | 2.17
  Aspartate aminotransferase (AST) (n=1013) | 2.07
  Absolute Neutrophil Count (n=1004) | 0.70
  Alkaline Phosphatase (n=1014) | 0.39
  Creatinine (n=1014) | 0.49
  Gamma-glutamyl transpeptidase (GGT) (n=1014) | 4.73
  Hemoglobin (n=1005) | 0.20
  Hyperbilirubinemia (n=1013) | 1.28
  Hyperuricemia (n=1014) | 0.69
  Hypophosphatemia (n=1014) | 0.20
  Lipase (n=409) | 4.40
  Platelets (n=997) | 1.50
  Potassium (hyperkalemia) (n=1014) | 0.10
  Serum Amylase (n=1014) | 4.83
  Sodium (hypernatremia) (n=1014) | 0.10
  Triglycerides (n=1014) | 4.73

3. Primary Outcome: Percentage of Participants With Grade 4 Laboratory Abnormalities Without Regards to Baseline Abnormalities
Description: Laboratory abnormalities as defined by the Division of AIDS (DAIDS) toxicity grading scale: Grade 4, Very Severe = events which were unacceptable and intolerable or were irreversible or caused the participant to be in imminent danger of death.
Time Frame: Baseline up to Week 144
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 1014
percentage of participants
  ALT (n=1013) | 0.79
  AST (n=1013) | 0.39
  Absolute Neutrophil Count (n=1004) | 0.20
  Alkaline Phosphatase (n=1014) | 0.00
  Creatinine (n=1014) | 0.10
  GGT (n=1014) | 1.48
  Hemoglobin (n=1005) | 0.10
  Hyperbilirubinemia (n=1013) | 0.30
  Hyperuricemia (n=1014) | 0.10
  Hypophosphatemia (n=1014) | 0.00
  Lipase (n=409) | 1.22
  Platelets (n=997) | 0.30
  Potassium (hyperkalemia) (n=1014) | 0.20
  Serum Amylase (n=1014) | 0.30
  Sodium (hypernatremia) (n=1014) | 0.20
  Triglycerides (n=1014) | 1.97

4. Primary Outcome: Percentage of Participants With Acquired Immunodeficiency Syndrome (AIDS)-Defining Illnesses
Description: Treatment-emergent AIDS-defining opportunistic illnesses based on investigator classification guided by a predefined list of clinical Category C adverse events per Center for Disease Control (CDC) HIV Classification System. Includes events occurring up to 30 days after last dose of study drug.
Time Frame: Baseline up to Week 144
Population: Safety analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 1032
percentage of participants
  AIDS encephalopathy | 0.1
  Bone tuberculosis | 0.1
  Cytomegalovirus infection | 0.2
  Extrapulmonary tuberculosis | 0.1
  Meningitis cryptococcal | 0.1
  Meningitis tuberculous | 0.1
  Mycobacterium avium complex infection | 0.1
  Mycobacterium kansasii infection | 0.1
  Oesophageal candidiasis | 0.6
  Pancreatitis bacterial | 0.1
  Pneumocystis jiroveci pneumonia | 0.1
  Progressive multifocal leukoencephalopathy | 0.1
  Pulmonary tuberculosis | 0.5
  Toxoplasmosis | 0.1
  B-cell lymphoma | 0.1
  Hodgkin's disease | 0.1
  Kaposi's sarcoma | 0.2
  Encephalopathy | 0.1

5. Primary Outcome: Percentage of Participants With Possible Acquired Immunodeficiency Syndrome (AIDS) Related Infections and Malignancies by Baseline Viral Load
Time Frame: Baseline up to Week 144
Population: Safety analysis set. Data not analyzed; the number of possible AIDS-related infections and malignancies and limited data collection during the study in terms of baseline viral load were such that a summary of AIDS-related infections by this parameter was not clinically meaningful.
Arm/Group | Maraviroc
Number analyzed (Participants) | 0

6. Primary Outcome: Percentage of Participants With Possible Acquired Immunodeficiency Syndrome (AIDS) Related Infections and Malignancies by Baseline/Nadir CD4 Cell Counts
Time Frame: Baseline up to Week 144
Population: Safety analysis set. Data not analyzed; the number of possible AIDS-related infections and malignancies and limited data collection during the study in terms of baseline/nadir CD4 cell counts were such that a summary of AIDS-related infections by this parameter was not clinically meaningful.
Arm/Group | Maraviroc
Number analyzed (Participants) | 0

7. Primary Outcome: Percentage of Participants With Possible Acquired Immunodeficiency Syndrome (AIDS) Related Infections and Malignancies by Time on Therapy
Time Frame: Baseline up to Week 144
Population: Safety analysis set. Data not analyzed; the number of possible AIDS-related infections and malignancies and limited data collection during the study by time on therapy were such that a summary of AIDS-related infections by this parameter was not clinically meaningful.
Arm/Group | Maraviroc
Number analyzed (Participants) | 0

8. Primary Outcome: Percentage of Participants With All Causality Treatment-emergent Adverse (AEs) Events by Gender
Description: Treatment-emergent AEs by gender that occurred up to 30 days after the last dose of study medication.
Time Frame: Baseline up to Week 144
Population: Safety analysis set; n = number of participants evaluable for adverse events.
Measure: Number; unit: percentage of participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 1032
percentage of participants
  Male (n=827) | 69.6
  Female (n=205) | 73.7

9. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (AEs) by Race
Description: Treatment-emergent AEs by race that occurred up to 30 days after the last dose of study medication.
Time Frame: Baseline up to Week 144
Population: Safety analysis set; n = number of participants evaluable for adverse events.
Measure: Number; unit: percentage of participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 1032
percentage of participants
  White (n=817) | 68.5
  Black (n=106) | 67.9
  Asian (n=54) | 88.9
  Other Unspecified (n=55) | 85.5

10. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (AEs) by Age
Description: Treatment-emergent AEs by age that occurred up to 30 days after the last dose of study medication.
Time Frame: Baseline up to Week 144
Population: Safety analysis set; n = number of participants evaluable for adverse events.
Measure: Number; unit: percentage of participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 1032
percentage of participants
  <18 years (n=1) | 100.0
  18 to 44 years (n=515) | 71.7
  45 to 64 years (n=493) | 68.6
  >=65 years (n=23) | 82.6

11. Primary Outcome: Percentage of Participants With Treatment-emergent Averse Events (AEs) by Baseline Hepatitis B and Hepatitis C Virus Serology Status
Description: Treatment emergent AEs by hepatis B and hepatitis C serology status that occurred up to 30 days post last dose.
Time Frame: Baseline up to Week 144
Population: Safety analysis set; n = number of participants evaluable for adverse events. Abbreviations: HBV = hepatitis B virus, HBC = hepatitis C virus.
Measure: Number; unit: percentage of participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 1032
percentage of participants
  HBV: negative (n=897) | 71.3
  HBV: positive (n=60) | 65.0
  HBV: missing: (n=75) | 64.0
  HCV: negative (n=794) | 72.7
  HCV: positive (n=158) | 62.7
  HCV: missing (n=80) | 63.8

12. Secondary Outcome: Percentage of Participants With ≥0.5 log10 Reduction From Baseline in Human Immunodeficiency Virus 1 Ribonucleic Acid (HIV 1 RNA)
Description: Defined as HIV-1 RNA levels < 400 Copies/mL or at least 0.5 Log 10-decrease from baseline in HIV-1 RNA levels.
  Baseline value calculated as average of the screening and baseline values if both values were within 1 log10 difference.
Time Frame: Baseline up to Week 144
Population: Safety analysis set; n = number of participants contributing to summary statistic at given timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 1032
percentage of participants
  Day 2-7 (n=26) | 46.2
  Week 2 (n=226) | 93.8
  Week 4 (n=773) | 93
  Week 8 (n=761) | 93.2
  Week 12 (n=756) | 94
  Week 16 (n=155) | 87.7
  Week 20 (n=131) | 93.1
  Week 24 (n=557) | 91.9
  Week 32 (n=202) | 93.1
  Week 40 (n=227) | 91.2
  Week 48 (n=228) | 89
  Week 60 (n=160) | 90
  Week 72 (n=125) | 88
  Week 84 (n=79) | 84.8
  Week 96 (n=48) | 91.7
  Week 108 (n=18) | 100
  Week 120 (n=9) | 100
  Week 132 (n=4) | 100
  Week 144 (n=1) | 100

13. Secondary Outcome: Percentage of Participants With ≥1.0 log10 Reduction From Baseline in HIV 1 RNA
Description: Defined as HIV-1 RNA levels < 400 copies/mL or at least 1.0 Log 10-decrease from baseline in HIV-1 RNA levels. Baseline value calculated as average of the screening and baseline values if both values were within 1 log10 difference.
Time Frame: Baseline up to Week 144
Population: Safety analysis set; n = number of participants contributing to summary statistic at given timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 1032
percentage of participants
  Day 2-7 (n=26) | 30.8
  Week 2 (n=226) | 90.3
  Week 4 (n=773) | 90.2
  Week 8 (n=761) | 91.2
  Week 12 (n=756) | 91.3
  Week 16 (n=155) | 82.6
  Week 20 (n=131) | 89.3
  Week 24 (n=557) | 89
  Week 32 (n=202) | 90.1
  Week 40 (n=227) | 87.7
  Week 48 (n=228) | 86.4
  Week 60 (n=160) | 85.6
  Week 72 (n=125) | 83.2
  Week 84 (n=79) | 79.7
  Week 96 (n=48) | 85.4
  Week 108 (n=18) | 100
  Week 120 (n=9) | 100
  Week 132 (n=4) | 100
  Week 144 (n=1) | 100

14. Secondary Outcome: Percentage of Participants With HIV-1 RNA Levels Below the Limit of Quantification: <400 Copies/mL
Description: Limit of quantification defined as <400 copies/mL. Baseline value calculated as average of the screening and baseline values if both values were within 1 log 10 difference.
Time Frame: Baseline up to Week 144
Population: Safety analysis set; n = number of participants contributing to summary statistic at given timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 1032
percentage of participants
  Baseline (n=979) | 6.7
  Day 2-7 (n=26) | 3.8
  Week 2 (n=226) | 58.8
  Week 4 (n=773) | 72.7
  Week 8 (n=761) | 78.8
  Week 12 (n=756) | 82.5
  Week 16 (n=155) | 75.5
  Week 20 (n=131) | 83.2
  Week 24 (n=557) | 84.4
  Week 32 (n=202) | 83.7
  Week 40 (n=227) | 81.1
  Week 48 (n=228) | 80.7
  Week 60 (n=160) | 78.1
  Week 72 (n=125) | 72.8
  Week 84 (n=79) | 74.7
  Week 96 (n=48) | 75.0
  Week 108 (n=18) | 88.9
  Week 120 (n=9) | 77.8
  Week 132 (n=4) | 100
  Week 144 (n=1) | 100

15. Secondary Outcome: Percentage of Participants With HIV-1 RNA Levels Below the Limit of Quantification: <50 Copies/mL
Description: Limit of quantification defined as <50 copies/mL. Baseline value calculated as average of the screening and baseline values if both values were within 1 log 10 difference.
Time Frame: Baseline up to Week 144
Population: Safety analysis set; n = number of participants contributing to summary statistic at given timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 1032
percentage of participants
  Baseline (n=979) | 1.7
  Day 2-7 (n=26) | 0.0
  Week 2 (n=226) | 19.9
  Week 4 (n=773) | 30.1
  Week 8 (n=761) | 43.1
  Week 12 (n=756) | 45.8
  Week 16 (n=155) | 37.4
  Week 20 (n=131) | 42.7
  Week 24 (n=557) | 55.8
  Week 32 (n=202) | 57.4
  Week 40 (n=227) | 54.6
  Week 48 (n=228) | 54.8
  Week 60 (n=160) | 51.9
  Week 72 (n=125) | 49.6
  Week 84 (n=79) | 55.7
  Week 96 (n=48) | 54.2
  Week 108 (n=18) | 77.8
  Week 120 (n=9) | 44.4
  Week 132 (n=4) | 75.0
  Week 144 (n=1) | 100

16. Secondary Outcome: Change From Baseline in CD4 Cell Count
Description: Change from baseline in cluster of differentiation 4 helper T cells (CD4) cell count. If baseline value was not available, it was taken from immediate preceding non-missing value.
Time Frame: Baseline up to Week 144
Population: Safety analysis set; n = number of participants contributing to summary statistic at given timepoint.
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Maraviroc
Number analyzed (Participants) | 1032
cells/uL
  Day 2-7 (n=6) | 28.5 (76.18)
  Week 2 (n=213) | 49.7 (93.15)
  Week 4 (n=762) | 68.9 (124.31)
  Week 8 (n=739) | 94.5 (122.94)
  Week 12 (n=738) | 95.7 (124.42)
  Week 16 (n=149) | 85.9 (124.37)
  Week 20 (n=130) | 106.6 (112.26)
  Week 24 (n=552) | 127.8 (139.42)
  Week 32 (n=197) | 124.1 (150.44)
  Week 40 (n=232) | 129.2 (144.31)
  Week 48 (n=222) | 140.5 (154.46)
  Week 60 (n=161) | 134.0 (151.52)
  Week 72 (n=124) | 147.0 (160.92)
  Week 84 (n=72) | 141.1 (147.55)
  Week 96 (n=50) | 160.3 (160.78)
  Week 108 (n=19) | 242.9 (167.06)
  Week 120 (n=8) | 117.9 (203.49)
  Week 132 (n=4) | 179.0 (109.94)
  Week 144 (n=1) | 93.0 (NA) — No standard deviation for 1 participant analyzed.

17. Secondary Outcome: Change From Baseline in CD4 Cell Count Percent
Description: Change from baseline in CD4 cell count percent . If baseline value was not available, it was taken from immediate preceding non-missing value.
Time Frame: Baseline up to Week 144
Population: Safety analysis set; n = number of participants contributing to summary statistic at given timepoint.
Measure: Mean (Standard Deviation); unit: percentage of lymphocytes
Arm/Group | Maraviroc
Number analyzed (Participants) | 1032
percentage of lymphocytes
  Days 2-7 (n=6) | -1.3 (1.56)
  Week 2 (n=206) | 1.8 (3.79)
  Week 4 (n=733) | 1.6 (4.84)
  Week 8 (n=722) | 1.4 (6.12)
  Week 12 (n=708) | 1.6 (5.45)
  Week 16 (n=141) | 1.9 (4.63)
  Week 20 (n=125) | 2.2 (6.17)
  Week 24 (n=531) | 2.8 (4.55)
  Week 32 (n=191) | 3.2 (5.38)
  Week 40 (n=218) | 3.7 (4.97)
  Week 48 (n=210) | 3.5 (5.87)
  Week 60 (n=148) | 4.5 (6.10)
  Week 72 (n=116) | 5.0 (6.33)
  Week 84 (n=64) | 5.7 (6.73)
  Week 96 (n=41) | 3.9 (6.36)
  Week 108 (n=19) | 6.3 (6.86)
  Week 120 (n=7) | 5.7 (9.07)
  Week 132 (n=4) | 8.5 (8.35)
  Week 144 (n=1) | 1.0 (0.0)

18. Secondary Outcome: Change From Baseline in CD8 Cell Count
Description: Change from baseline in cluster of differentiation 8 suppressor T cells (CD8) cell count. If baseline value was not available, it was taken from immediate preceding non-missing value.
Time Frame: Baseline up to Week 144
Population: Safety analysis set; n = number of participants contributing to summary statistic at given timepoint.
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Maraviroc
Number analyzed (Participants) | 1032
cells/uL
  Day 2-7 (n=6) | 268.5 (262.50)
  Week 2 (n=201) | 78.2 (343.85)
  Week 4 (n=701) | 205.6 (509.70)
  Week 8 (n=692) | 345.6 (599.98)
  Week 12 (n=696) | 309.4 (578.91)
  Week 16 (n=129) | 259.6 (430.78)
  Week 20 (n=119) | 325.2 (621.46)
  Week 24 (n=523) | 251.3 (498.85)
  Week 32 (n=185) | 185.2 (484.74)
  Week 40 (n=222) | 160.9 (471.99)
  Week 48 (n=214) | 153.2 (464.73)
  Week 60 (n=157) | 76.9 (467.64)
  Week 72 (n=120) | 68.7 (502.73)
  Week 84 (n=70) | -11.6 (548.85)
  Week 96 (n=45) | 56.6 (403.10)
  Week 108 (n=19) | 147.5 (600.55)
  Week 120 (n=8) | -135.1 (517.02)
  Week 132 (n=4) | -363.3 (882.30)
  Week 144 (n=1) | 642.0 (0.0)

19. Secondary Outcome: Change From Baseline in CD8 Cell Count Percent
Description: Change from baseline in CD8 cell count percent . If baseline value was not available, it was taken from immediate preceding non-missing value.
Time Frame: Baseline up to Week 144
Population: Safety analysis set; n = number of participants contributing to summary statistic at given timepoint.
Measure: Mean (Standard Deviation); unit: percentage of lymphocytes
Arm/Group | Maraviroc
Number analyzed (Participants) | 1032
percentage of lymphocytes
  Day 2-7 (n=6) | 3.0 (3.42)
  Week 2 (n=197) | -1.5 (7.68)
  Week 4 (n=689) | -0.3 (8.08)
  Week 8 (n=683) | 0.4 (9.62)
  Week 12 (n=675) | -0.9 (9.95)
  Week 16 (n=125) | 0.7 (8.66)
  Week 20 (n=115) | -0.7 (10.08)
  Week 24 (n=510) | -3.2 (8.92)
  Week 32 (n=184) | -4.0 (9.09)
  Week 40 (n=215) | -4.5 (8.90)
  Week 48 (n=202) | -5.1 (10.63)
  Week 60 (n=146) | -5.0 (11.90)
  Week 72 (n=113) | -6.2 (9.87)
  Week 84 (n=64) | -8.2 (15.52)
  Week 96 (n=40) | -9.5 (10.18)
  Week 108 (n=19) | -14.5 (9.99)
  Week 120 (n=6) | -14.5 (13.41)
  Week 132 (n=4) | -16.8 (12.89)
  Week 144 (n=1) | -2.0 (0.0)

20. Secondary Outcome: Median Time to Virologic Failure
Description: Computed as time from the first dose of study medication to the loss of virologic response. Virologic failure defined as: failure to achieve a reduction from baseline (BL) in HIV 1 RNA ≥ 0.5 log10 copies /mL by the second viral load determination (unless viral load was below the lower limit level of quantification [LLOQ]); or a ≥ 0.5 log10 increase from nadir in HIV 1 RNA after achieving a HIV 1 RNA reduction from BL >0.5 log10 copies/mL; or a HIV 1 RNA level of >1000 copies/mL after having achieved a HIV 1 RNA level below LLOQ.
Time Frame: Day 1 up to Week 144
Population: Safety analysis set. N = number of participants with virologic failure. For the calculation of the time to virologic failure, any visits with no data were excluded. Participants who were not virologic failures were censored at the last available observation.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Maraviroc
Number analyzed (Participants) | 192
days | 86.5 [58.0 to 169.0]
Statistical Analysis 1: Comparison: Maraviroc; Test type: Superiority or Other; 75th percentile (median) = 169.0, 95% CI 2-sided [135.0 to 178.0]
Statistical Analysis 2: Comparison: Maraviroc; Test type: Superiority or Other; 50th percentile (median) = 86.5, 95% CI 2-sided [82.0 to 92.0]
Statistical Analysis 3: Comparison: Maraviroc; Test type: Superiority or Other; 25th percentile (median) = 58.0, 95% CI 2-sided [57.0 to 62.0]

21. Secondary Outcome: Percentage of Participants With Changes in HIV-1 RNA Level in Participants Meeting the Definition of Virologic Failure
Description: Reasons for virologic failure: A) failure to achieve a reduction in HIV-1 RNA>=0.5 log10 copies/ml from baseline (BL) by second viral load determination (unless below level of quantification [LOQ]); B) >=0.5 log10 increase from nadir in HIV-1 RNA after achieving an HIV-1 RNA reduction from BL >0.5 log10 copies/ml ; C) HIV-1 RNA >1000 copies/ml after having achieved an HIV-1 RNA below LOQ.
Time Frame: Baseline up to Week 144
Population: Safety analysis set; N = number of participants with virologic failure.
Measure: Number; unit: percentage of participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 192
percentage of participants
  Reduction in HIV-1 RNA<0.5 log10 copies/ml | 43.75
  >=0.5 log10 increase from nadir in HIV-1 RNA | 31.77
  HIV-1 RNA >1000 copies/ml | 18.75
  Reduction <0.5 log10 + HIV-1 RNA >1000 copies/ml | 3.13
  >=0.5 log10 increase from nadir + HIV-1 RNA >1000 | 2.60

22. Secondary Outcome: Percentage of Participants With Change in Chemokine Co-receptor Tropism From Screening to Time of Virologic Failure
Description: Tropism status (CCR5 [R5], CXCR4 [X4], Dual Mixed [DM], or Non-reportable [NR]) at Screening (Scr) and time of virologic failure (V fail). Virologic failure defined as: failure to achieve a reduction from baseline (BL) in HIV 1 RNA ≥0.5 log10 copies/mL by second viral load determination (unless viral load was below lower limit level of quantification [LLOQ]); or a ≥ 0.5 log10 increase from nadir in HIV 1 RNA after achieving HIV 1 RNA reduction from BL >0.5 log10 copies/mL; or a HIV 1 RNA level of >1000 copies/mL after having achieved a HIV 1 RNA level below LLOQ.
Time Frame: Screening up to Week 144
Population: Safety analysis set; N = participants with virologic failure (VF). Abbreviations: Scr = screening, R5 = CCR5 tropic HIV-1, X4=CXCR4 tropic HIV-1, DM = dual mixed, NR = non-reportable, Missing = participants with VF who did not have tropism result within specified screening period (Scr missing: -42 days to Day 0) or at the time of VF.
Measure: Number; unit: percentage of participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 192
percentage of participants
  Scr: Missing; V fail: R5 | 5.73
  Scr: Missing; V fail: X4 | 0.52
  Scr: Missing; V fail: DM | 1.04
  Scr: Missing; V fail: NR | 7.29
  Scr: Missing; V fail: Missing | 1.56
  Scr: NR; V fail: R5 | 0.52
  Scr: R5; V fail: R5 | 31.25
  Scr: R5; V fail: X4 | 4.17
  Scr: R5; V fail: DM | 18.75
  Scr: R5; V fail: NR | 22.92
  Scr: R5; V fail: Missing | 6.25

23. Secondary Outcome: Number of Participants With Reduced Maraviroc Susceptibility as Defined by Change From Baseline to Time of Virologic Failure in Inhibitory Concentration of 50% (IC 50) and Presence of Plateau
Description: Resistance to maravroc in viruses from participants failing therapy with R5 virus was investigated using the in vitro phenotypic (drug susceptibility) assay. The number of participants who failed with R5 virus were assessed successfully for maraviroc susceptibility at Baseline and Last on--treatment (Week 144). Samples were analyzed for change from Baseline to time of virologic failure in IC 50 and presence of plateau. A maximal percent inhibition (MPI) <95% established as a plateau in inhibition at high concentrations of maraviroc was used to identify viruses which had reduced phenotypic susceptibility to maraviroc.
Time Frame: Baseline up to Week 144
Population: Safety analysis set. Here, "number of participants analyzed" signifies those participants who were assessed for maraviroc susceptibility.
Measure: Number; unit: participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 26
participants | 14

24. Secondary Outcome: Number of Participants With Emergence of Resistance to Maraviroc as Defined by Genotypic Changes in the V3 Loop of Glycoprotein 120 (gp 120)
Description: Virus from participants who experienced virologic failure was analyzed for resistance to maraviroc. Resistance testing was performed on archived samples of participants which were available pre--treatment at time of virologic failure. For participants who met definition of virologic failure during the trial, the sequencing of the V3 loop of HIV--1 viral envelope gp 120 was evaluated to identify any amino acid changes concomitant with decreased susceptibility to maraviroc.
Time Frame: Baseline up to Week 144
Population: Safety analysis set. Here, "number of participants analyzed" signifies those participants who were assessed for genotypic changes in the V3 Loop of glycoprotein 120 (gp 120).
Measure: Number; unit: participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 13
participants | NA — Data was not evaluable because of lack of any distinct mutational pattern for resistance in analyzed participants.

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Maraviroc
Serious Adverse Events (participants affected / at risk) | 139/1032
Other Adverse Events (participants affected / at risk) | 700/1032
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Maraviroc (N=1032)
Anaemia (Blood and lymphatic system disorders) | 5
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Acute coronary syndrome (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Congestive cardiomyopathy (Cardiac disorders) | 1
Left ventricular failure (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 3
Palpitations (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 2
Vision blurred (Eye disorders) | 1
Visual impairment (Eye disorders) | 2
Vitreous floaters (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Anal fissure (Gastrointestinal disorders) | 1
Anogenital dysplasia (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 7
Food poisoning (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Oesophagitis (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Peptic ulcer (Gastrointestinal disorders) | 1
Rectal polyp (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Chest pain (General disorders) | 7
Chills (General disorders) | 1
Drug interaction (General disorders) | 1
Gait disturbance (General disorders) | 1
General physical health deterioration (General disorders) | 3
Hyperthermia (General disorders) | 1
Pyrexia (General disorders) | 10
Bile duct stone (Hepatobiliary disorders) | 1
Cytolytic hepatitis (Hepatobiliary disorders) | 4
Hepatic failure (Hepatobiliary disorders) | 1
Hepatitis cholestatic (Hepatobiliary disorders) | 1
Hepatotoxicity (Hepatobiliary disorders) | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 2
Immune reconstitution syndrome (Immune system disorders) | 1
AIDS encephalopathy (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 2
Bone tuberculosis (Infections and infestations) | 1
Bronchitis fungal (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Dengue fever (Infections and infestations) | 1
Dermo-hypodermitis (Infections and infestations) | 1
Dysentery (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 2
Extradural abscess (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
HIV infection (Infections and infestations) | 1
Hepatitis B (Infections and infestations) | 2
Herpes zoster (Infections and infestations) | 3
Influenza (Infections and infestations) | 1
Intervertebral discitis (Infections and infestations) | 1
Leptospirosis (Infections and infestations) | 1
Lower respiratory tract infection bacterial (Infections and infestations) | 1
Mastoiditis (Infections and infestations) | 1
Meningitis cryptococcal (Infections and infestations) | 1
Meningitis tuberculous (Infections and infestations) | 1
Mycobacterium avium complex infection (Infections and infestations) | 1
Mycobacterium kansasii infection (Infections and infestations) | 1
Pancreatitis bacterial (Infections and infestations) | 1
Pneumococcal sepsis (Infections and infestations) | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 11
Pneumonia bacterial (Infections and infestations) | 2
Pneumonia legionella (Infections and infestations) | 2
Pseudomonas infection (Infections and infestations) | 1
Pulmonary tuberculosis (Infections and infestations) | 3
Respiratory tract infection (Infections and infestations) | 1
Respiratory tract infection bacterial (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Septic shock (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 2
Staphylococcal bacteraemia (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 4
Ankle fracture (Injury, poisoning and procedural complications) | 1
Drug toxicity (Injury, poisoning and procedural complications) | 3
Femur fracture (Injury, poisoning and procedural complications) | 1
Joint injury (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Blood alkaline phosphatase increased (Investigations) | 2
Blood creatine phosphokinase increased (Investigations) | 2
Blood glucose increased (Investigations) | 1
Clostridium test positive (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Weight decreased (Investigations) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Diabetic foot (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carcinoma in situ of penis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Brain oedema (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 3
Disturbance in attention (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Anxiety disorder (Psychiatric disorders) | 1
Completed suicide (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Hallucination, auditory (Psychiatric disorders) | 1
Homicidal ideation (Psychiatric disorders) | 1
Major depression (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 2
Renal failure (Renal and urinary disorders) | 3
Renal failure acute (Renal and urinary disorders) | 4
Urinary bladder polyp (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1
Coronary artery bypass (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 2
Hypertensive crisis (Vascular disorders) | 2
Orthostatic hypotension (Vascular disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Maraviroc (N=1032)
Agranulocytosis (Blood and lymphatic system disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 18
Bone marrow failure (Blood and lymphatic system disorders) | 1
Eosinophilia (Blood and lymphatic system disorders) | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 18
Microcytic anaemia (Blood and lymphatic system disorders) | 2
Microcytosis (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Polycythaemia (Blood and lymphatic system disorders) | 1
Splenomegaly (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Angina pectoris (Cardiac disorders) | 3
Cardiac failure congestive (Cardiac disorders) | 2
Cyanosis (Cardiac disorders) | 1
Extrasystoles (Cardiac disorders) | 1
Hyperdynamic left ventricle (Cardiac disorders) | 1
Left atrial dilatation (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 3
Pericardial effusion (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 5
Accessory spleen (Congenital, familial and genetic disorders) | 1
Dysmorphism (Congenital, familial and genetic disorders) | 1
Preauricular cyst (Congenital, familial and genetic disorders) | 1
Cerumen impaction (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 7
Tinnitus (Ear and labyrinth disorders) | 4
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 12
Goitre (Endocrine disorders) | 2
Hypogonadism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1
Blepharitis (Eye disorders) | 3
Blindness unilateral (Eye disorders) | 1
Cataract (Eye disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 10
Conjunctivitis allergic (Eye disorders) | 2
Dry eye (Eye disorders) | 1
Exophthalmos (Eye disorders) | 1
Eye irritation (Eye disorders) | 2
Eye swelling (Eye disorders) | 1
Foreign body sensation in eyes (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Metamorphopsia (Eye disorders) | 1
Ocular icterus (Eye disorders) | 1
Punctate keratitis (Eye disorders) | 1
Pupils unequal (Eye disorders) | 1
Uveitis (Eye disorders) | 1
Vision blurred (Eye disorders) | 7
Visual acuity reduced (Eye disorders) | 3
Visual impairment (Eye disorders) | 5
Vitreous detachment (Eye disorders) | 1
Vitreous floaters (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 12
Abdominal pain (Gastrointestinal disorders) | 20
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 14
Abdominal tenderness (Gastrointestinal disorders) | 1
Anal fistula (Gastrointestinal disorders) | 1
Anal polyp (Gastrointestinal disorders) | 1
Anal ulcer (Gastrointestinal disorders) | 1
Anogenital dysplasia (Gastrointestinal disorders) | 1
Anorectal discomfort (Gastrointestinal disorders) | 1
Anorectal disorder (Gastrointestinal disorders) | 4
Aphthous stomatitis (Gastrointestinal disorders) | 5
Cheilitis (Gastrointestinal disorders) | 5
Colitis (Gastrointestinal disorders) | 2
Colitis ulcerative (Gastrointestinal disorders) | 1
Colonic polyp (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 35
Defaecation urgency (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 94
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 6
Dyspepsia (Gastrointestinal disorders) | 13
Dysphagia (Gastrointestinal disorders) | 6
Eructation (Gastrointestinal disorders) | 1
Faecal incontinence (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 14
Food poisoning (Gastrointestinal disorders) | 1
Gastric disorder (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 10
Gastrointestinal disorder (Gastrointestinal disorders) | 5
Gastrointestinal pain (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9
Gingivitis (Gastrointestinal disorders) | 5
Glossitis (Gastrointestinal disorders) | 2
Haematochezia (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 13
Hyperchlorhydria (Gastrointestinal disorders) | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 60
Odynophagia (Gastrointestinal disorders) | 3
Oesophagitis (Gastrointestinal disorders) | 3
Oral discomfort (Gastrointestinal disorders) | 1
Oral disorder (Gastrointestinal disorders) | 1
Oral lichen planus (Gastrointestinal disorders) | 1
Painful defaecation (Gastrointestinal disorders) | 2
Paraesthesia oral (Gastrointestinal disorders) | 1
Parotid gland enlargement (Gastrointestinal disorders) | 2
Periodontitis (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 6
Salivary gland cyst (Gastrointestinal disorders) | 1
Tongue discolouration (Gastrointestinal disorders) | 1
Tongue disorder (Gastrointestinal disorders) | 1
Tongue ulceration (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 2
Umbilical hernia (Gastrointestinal disorders) | 2
Uvulitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 34
Adverse drug reaction (General disorders) | 1
Asthenia (General disorders) | 21
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 9
Chills (General disorders) | 5
Crepitations (General disorders) | 1
Facial pain (General disorders) | 1
Fat tissue increased (General disorders) | 1
Fatigue (General disorders) | 24
Feeling hot (General disorders) | 1
Feeling jittery (General disorders) | 1
Influenza like illness (General disorders) | 14
Injection site nodule (General disorders) | 1
Injection site reaction (General disorders) | 8
Injection site swelling (General disorders) | 1
Irritability (General disorders) | 1
Local swelling (General disorders) | 2
Malaise (General disorders) | 4
Mucosal inflammation (General disorders) | 1
Necrosis (General disorders) | 1
Nodule (General disorders) | 3
Oedema (General disorders) | 3
Oedema peripheral (General disorders) | 12
Pain (General disorders) | 15
Pyrexia (General disorders) | 50
Thirst (General disorders) | 1
Ulcer (General disorders) | 3
Cholelithiasis (Hepatobiliary disorders) | 1
Cholestasis (Hepatobiliary disorders) | 1
Cytolytic hepatitis (Hepatobiliary disorders) | 7
Hepatic steatosis (Hepatobiliary disorders) | 2
Hepatitis acute (Hepatobiliary disorders) | 1
Hepatomegaly (Hepatobiliary disorders) | 8
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 4
Liver disorder (Hepatobiliary disorders) | 2
Allergy to arthropod bite (Immune system disorders) | 1
Drug hypersensitivity (Immune system disorders) | 3
Food allergy (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 2
Immune reconstitution syndrome (Immune system disorders) | 3
Seasonal allergy (Immune system disorders) | 1
Abscess (Infections and infestations) | 1
Abscess limb (Infections and infestations) | 1
Acarodermatitis (Infections and infestations) | 2
Acute sinusitis (Infections and infestations) | 2
Amoebic dysentery (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 2
Anal fungal infection (Infections and infestations) | 1
Anogenital warts (Infections and infestations) | 6
Body tinea (Infections and infestations) | 2
Bronchiolitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 67
Bronchitis bacterial (Infections and infestations) | 1
Campylobacter intestinal infection (Infections and infestations) | 1
Candidiasis (Infections and infestations) | 5
Cellulitis (Infections and infestations) | 8
Chronic sinusitis (Infections and infestations) | 3
Conjunctivitis viral (Infections and infestations) | 1
Cystitis (Infections and infestations) | 5
Cytomegalovirus infection (Infections and infestations) | 2
Dermo-hypodermitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Ear infection (Infections and infestations) | 5
Extrapulmonary tuberculosis (Infections and infestations) | 1
Eye infection (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 6
Fungal infection (Infections and infestations) | 3
Fungal skin infection (Infections and infestations) | 5
Furuncle (Infections and infestations) | 3
Gastroenteritis (Infections and infestations) | 17
Gastroenteritis viral (Infections and infestations) | 2
Gastrointestinal infection (Infections and infestations) | 4
Gastrointestinal viral infection (Infections and infestations) | 1
Genital abscess (Infections and infestations) | 1
Genital herpes (Infections and infestations) | 12
Genital infection fungal (Infections and infestations) | 3
Genitourinary chlamydia infection (Infections and infestations) | 1
Gingival infection (Infections and infestations) | 1
Gonorrhoea (Infections and infestations) | 1
Haematoma infection (Infections and infestations) | 1
Haemophilus infection (Infections and infestations) | 1
Helicobacter gastritis (Infections and infestations) | 2
Hepatitis A (Infections and infestations) | 1
Hepatitis B (Infections and infestations) | 3
Hepatitis C (Infections and infestations) | 6
Herpes simplex (Infections and infestations) | 14
Herpes virus infection (Infections and infestations) | 10
Herpes zoster (Infections and infestations) | 18
Hordeolum (Infections and infestations) | 1
Impetigo (Infections and infestations) | 2
Infected bites (Infections and infestations) | 1
Infection (Infections and infestations) | 3
Infestation (Infections and infestations) | 1
Influenza (Infections and infestations) | 29
Laryngitis (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 5
Lymphangitis (Infections and infestations) | 1
Mastitis (Infections and infestations) | 1
Mastoiditis (Infections and infestations) | 1
Meningitis aseptic (Infections and infestations) | 1
Molluscum contagiosum (Infections and infestations) | 2
Mycotic corneal ulcer (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 41
Oesophageal candidiasis (Infections and infestations) | 6
Onychomycosis (Infections and infestations) | 6
Oral candidiasis (Infections and infestations) | 28
Oral fungal infection (Infections and infestations) | 3
Oral hairy leukoplakia (Infections and infestations) | 3
Oral herpes (Infections and infestations) | 13
Oral infection (Infections and infestations) | 1
Orchitis (Infections and infestations) | 2
Otitis externa (Infections and infestations) | 3
Otitis media (Infections and infestations) | 7
Otitis media acute (Infections and infestations) | 1
Papilloma viral infection (Infections and infestations) | 4
Paronychia (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 22
Pneumococcal infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 6
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1
Prostatitis Escherichia coli (Infections and infestations) | 1
Pulmonary tuberculosis (Infections and infestations) | 2
Purulent discharge (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 2
Rash pustular (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 5
Respiratory tract infection viral (Infections and infestations) | 2
Rhinitis (Infections and infestations) | 13
Scrotal infection (Infections and infestations) | 1
Secondary syphilis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Shigella infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 28
Skin infection (Infections and infestations) | 3
Staphylococcal infection (Infections and infestations) | 3
Staphylococcal skin infection (Infections and infestations) | 1
Syphilis (Infections and infestations) | 7
Tinea cruris (Infections and infestations) | 3
Tinea infection (Infections and infestations) | 3
Tinea pedis (Infections and infestations) | 5
Tinea versicolour (Infections and infestations) | 2
Tooth abscess (Infections and infestations) | 3
Tooth infection (Infections and infestations) | 4
Toxoplasmosis (Infections and infestations) | 1
Tracheitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 41
Urethritis (Infections and infestations) | 2
Urethritis gonococcal (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 17
Urinary tract infection bacterial (Infections and infestations) | 1
Urinary tract infection enterococcal (Infections and infestations) | 1
Urinary tract infection fungal (Infections and infestations) | 1
Viral infection (Infections and infestations) | 6
Viral pharyngitis (Infections and infestations) | 1
Viral sinusitis (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 2
Vulvovaginal candidiasis (Infections and infestations) | 4
Wound infection (Infections and infestations) | 1
Animal bite (Injury, poisoning and procedural complications) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 3
Bone fissure (Injury, poisoning and procedural complications) | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 3
Epicondylitis (Injury, poisoning and procedural complications) | 2
Excoriation (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 3
Foot fracture (Injury, poisoning and procedural complications) | 3
Foreign body in eye (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Joint injury (Injury, poisoning and procedural complications) | 3
Joint sprain (Injury, poisoning and procedural complications) | 4
Ligament rupture (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 2
Muscle strain (Injury, poisoning and procedural complications) | 3
Overdose (Injury, poisoning and procedural complications) | 2
Periorbital haematoma (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Skeletal injury (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 2
Sunburn (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 13
Aspartate aminotransferase abnormal (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 9
Blood alkaline phosphatase (Investigations) | 1
Blood amylase increased (Investigations) | 11
Blood cholesterol increased (Investigations) | 2
Blood creatine increased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 8
Blood creatinine increased (Investigations) | 4
Blood glucose abnormal (Investigations) | 1
Blood glucose increased (Investigations) | 4
Blood iron decreased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Blood phosphorus decreased (Investigations) | 1
Blood pressure increased (Investigations) | 2
Blood sodium increased (Investigations) | 1
Blood triglycerides increased (Investigations) | 6
Blood uric acid increased (Investigations) | 6
Blood urine present (Investigations) | 1
Body temperature increased (Investigations) | 1
Cardiac function test abnormal (Investigations) | 1
Cardiac murmur (Investigations) | 3
Carotid bruit (Investigations) | 1
Eosinophil count increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 12
Glycosylated haemoglobin increased (Investigations) | 1
Haemoglobin decreased (Investigations) | 2
Helicobacter test positive (Investigations) | 1
Hepatic enzyme increased (Investigations) | 2
Hepatitis B DNA increased (Investigations) | 1
Hepatitis B antibody positive (Investigations) | 1
Hepatitis B positive (Investigations) | 1
Hepatitis B surface antigen positive (Investigations) | 3
Lipase increased (Investigations) | 7
Liver function test abnormal (Investigations) | 2
Low density lipoprotein increased (Investigations) | 1
Lymph node palpable (Investigations) | 2
Murphy's sign positive (Investigations) | 1
Occult blood positive (Investigations) | 1
Physical examination (Investigations) | 2
Platelet count decreased (Investigations) | 2
Prostatic specific antigen increased (Investigations) | 1
Serum ferritin increased (Investigations) | 1
Transaminases increased (Investigations) | 6
Treponema test positive (Investigations) | 1
Urine output decreased (Investigations) | 1
Waist circumference increased (Investigations) | 1
Weight decreased (Investigations) | 12
Weight increased (Investigations) | 11
Cell death (Metabolism and nutrition disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 9
Dehydration (Metabolism and nutrition disorders) | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 2
Dyslipidaemia (Metabolism and nutrition disorders) | 2
Folate deficiency (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 2
Hyperamylasaemia (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 6
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 25
Hyperuricaemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Hypocholesterolaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 6
Hypovolaemia (Metabolism and nutrition disorders) | 1
Impaired fasting glucose (Metabolism and nutrition disorders) | 2
Increased appetite (Metabolism and nutrition disorders) | 2
Malnutrition (Metabolism and nutrition disorders) | 2
Metabolic syndrome (Metabolism and nutrition disorders) | 1
Selenium deficiency (Metabolism and nutrition disorders) | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2
Vitamin C deficiency (Metabolism and nutrition disorders) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 2
Zinc deficiency (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 34
Arthritis (Musculoskeletal and connective tissue disorders) | 3
Arthropathy (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 45
Bone disorder (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Bursa disorder (Musculoskeletal and connective tissue disorders) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1
Enthesopathy (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 3
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 20
Neck pain (Musculoskeletal and connective tissue disorders) | 6
Nodule on extremity (Musculoskeletal and connective tissue disorders) | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1
Tendon pain (Musculoskeletal and connective tissue disorders) | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 4
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1
Torticollis (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oral papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Penile wart (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Testicular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ageusia (Nervous system disorders) | 1
Amnesia (Nervous system disorders) | 4
Aphasia (Nervous system disorders) | 1
Ataxia (Nervous system disorders) | 1
Carpal tunnel syndrome (Nervous system disorders) | 1
Central nervous system lesion (Nervous system disorders) | 1
Cerebral atrophy (Nervous system disorders) | 1
Decreased vibratory sense (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 26
Dysaesthesia (Nervous system disorders) | 2
Dysarthria (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Facial palsy (Nervous system disorders) | 2
Headache (Nervous system disorders) | 66
Hyperaesthesia (Nervous system disorders) | 1
Hypersomnia (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 2
Memory impairment (Nervous system disorders) | 3
Migraine (Nervous system disorders) | 3
Muscle contractions involuntary (Nervous system disorders) | 2
Nerve root compression (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 14
Paraesthesia (Nervous system disorders) | 6
Presyncope (Nervous system disorders) | 1
Radiculopathy (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 6
Sensory disturbance (Nervous system disorders) | 1
Serotonin syndrome (Nervous system disorders) | 1
Sleep phase rhythm disturbance (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 3
Syncope (Nervous system disorders) | 1
Tension headache (Nervous system disorders) | 1
Abnormal dreams (Psychiatric disorders) | 4
Aggression (Psychiatric disorders) | 1
Agitation (Psychiatric disorders) | 3
Anxiety (Psychiatric disorders) | 23
Bipolar I disorder (Psychiatric disorders) | 1
Bulimia nervosa (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 3
Depressed mood (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 20
Disorientation (Psychiatric disorders) | 1
Dysphoria (Psychiatric disorders) | 1
Euphoric mood (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Hallucination, auditory (Psychiatric disorders) | 1
Initial insomnia (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 32
Libido decreased (Psychiatric disorders) | 3
Libido disorder (Psychiatric disorders) | 1
Mental disorder (Psychiatric disorders) | 1
Mood altered (Psychiatric disorders) | 1
Nervousness (Psychiatric disorders) | 2
Sleep disorder (Psychiatric disorders) | 4
Stereotypy (Psychiatric disorders) | 1
Stress (Psychiatric disorders) | 2
Thinking abnormal (Psychiatric disorders) | 1
Tic (Psychiatric disorders) | 1
Withdrawal syndrome (Psychiatric disorders) | 1
Bladder disorder (Renal and urinary disorders) | 1
Calculus bladder (Renal and urinary disorders) | 1
Calculus ureteric (Renal and urinary disorders) | 1
Chromaturia (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 9
Haematuria (Renal and urinary disorders) | 4
Microalbuminuria (Renal and urinary disorders) | 1
Micturition disorder (Renal and urinary disorders) | 1
Micturition urgency (Renal and urinary disorders) | 1
Nephritis (Renal and urinary disorders) | 1
Nephroangiosclerosis (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 3
Nephropathy (Renal and urinary disorders) | 1
Nocturia (Renal and urinary disorders) | 2
Pollakiuria (Renal and urinary disorders) | 5
Polyuria (Renal and urinary disorders) | 3
Pyuria (Renal and urinary disorders) | 1
Renal cyst (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 4
Renal failure acute (Renal and urinary disorders) | 2
Renal impairment (Renal and urinary disorders) | 1
Renal pain (Renal and urinary disorders) | 1
Ureteral disorder (Renal and urinary disorders) | 1
Urinary hesitation (Renal and urinary disorders) | 3
Urinary incontinence (Renal and urinary disorders) | 3
Urinary tract disorder (Renal and urinary disorders) | 1
Amenorrhoea (Reproductive system and breast disorders) | 2
Balanitis (Reproductive system and breast disorders) | 2
Bartholin's cyst (Reproductive system and breast disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2
Breast cyst (Reproductive system and breast disorders) | 1
Breast pain (Reproductive system and breast disorders) | 2
Cervical polyp (Reproductive system and breast disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 10
Galactorrhoea (Reproductive system and breast disorders) | 1
Genital lesion (Reproductive system and breast disorders) | 1
Genital ulceration (Reproductive system and breast disorders) | 1
Gynaecomastia (Reproductive system and breast disorders) | 3
Metrorrhagia (Reproductive system and breast disorders) | 1
Oedema genital (Reproductive system and breast disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 2
Premenstrual syndrome (Reproductive system and breast disorders) | 1
Prostatic pain (Reproductive system and breast disorders) | 1
Prostatism (Reproductive system and breast disorders) | 2
Prostatitis (Reproductive system and breast disorders) | 7
Pruritus genital (Reproductive system and breast disorders) | 1
Retrograde ejaculation (Reproductive system and breast disorders) | 1
Scrotal ulcer (Reproductive system and breast disorders) | 1
Testicular pain (Reproductive system and breast disorders) | 1
Testicular swelling (Reproductive system and breast disorders) | 2
Uterine cyst (Reproductive system and breast disorders) | 1
Vaginal discharge (Reproductive system and breast disorders) | 1
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 6
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 47
Cyanosis central (Respiratory, thoracic and mediastinal disorders) | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 6
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 7
Rales (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 6
Rhinitis seasonal (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 10
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 2
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Tonsillar ulcer (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 4
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 6
Dandruff (Skin and subcutaneous tissue disorders) | 3
Dermal cyst (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 9
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2
Dermatosis (Skin and subcutaneous tissue disorders) | 2
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 9
Eczema (Skin and subcutaneous tissue disorders) | 4
Eosinophilic pustular folliculitis (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 4
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Facial wasting (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 1
Lichen planus (Skin and subcutaneous tissue disorders) | 1
Lipoatrophy (Skin and subcutaneous tissue disorders) | 2
Lipodystrophy acquired (Skin and subcutaneous tissue disorders) | 7
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 2
Night sweats (Skin and subcutaneous tissue disorders) | 7
Onychoclasis (Skin and subcutaneous tissue disorders) | 2
Penile ulceration (Skin and subcutaneous tissue disorders) | 1
Polymorphic light eruption (Skin and subcutaneous tissue disorders) | 1
Prurigo (Skin and subcutaneous tissue disorders) | 8
Pruritus (Skin and subcutaneous tissue disorders) | 22
Psoriasis (Skin and subcutaneous tissue disorders) | 4
Purpura (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 44
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Rash macular (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Rash papular (Skin and subcutaneous tissue disorders) | 6
Rash pruritic (Skin and subcutaneous tissue disorders) | 2
Rash vesicular (Skin and subcutaneous tissue disorders) | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 6
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2
Skin fibrosis (Skin and subcutaneous tissue disorders) | 1
Skin fragility (Skin and subcutaneous tissue disorders) | 1
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1
Skin induration (Skin and subcutaneous tissue disorders) | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 6
Skin nodule (Skin and subcutaneous tissue disorders) | 6
Skin reaction (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 3
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 4
Swelling face (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 3
Alcohol use (Social circumstances) | 1
Circumcision (Surgical and medical procedures) | 1
Dental implantation (Surgical and medical procedures) | 1
Prophylaxis (Surgical and medical procedures) | 1
Tooth extraction (Surgical and medical procedures) | 1
Wart excision (Surgical and medical procedures) | 1
Aortic stenosis (Vascular disorders) | 1
Flushing (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 1
Hot flush (Vascular disorders) | 2
Hypertension (Vascular disorders) | 22
Hypertensive crisis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 5
Pallor (Vascular disorders) | 1
Phlebitis (Vascular disorders) | 1
Thrombophlebitis (Vascular disorders) | 1
Venoocclusive disease (Vascular disorders) | 1
Venous insufficiency (Vascular disorders) | 3
Venous thrombosis (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Viral loads were not available for subjects uniformly as this expanded access study followed local country guidelines and practices that could vary significantly between countries, and testing frequency may have been affected by insurance status.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.